CLINICAL TRIAL: NCT06454279
Title: Effects of Cognitive Motor Dual Task Versus Task Specific Training on Cognition and Motor Functioning in Stroke Patients
Brief Title: Cognitive Motor Dual Task Versus Task Specific Training on Cognition and Motor Functioning in Stroke Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/MS-PT/018 Qudsia Hafeez
Record Dates: First submitted 2024-06-06; First posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Stroke
Keywords: Cognition, Motor Functioning, Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dual Task Training (Experimental): Dual task exercises for example Crossing over the obstacles placed on their path while answering simple questions "yes" or "no" Walking while bouncing the ball with spell the word like WORLD Picking up an object from the floor. Walking on straight line while Calculation. Tandem walk while counting money
  Interventions: Other: Dual Task Training
- Task Specific Training (Experimental): Picking up the card, Picking up the right color, Box and block activity, Picking up different shapes, Gait training, Sit/ standing marching.
  Interventions: Other: Task Specific Training

INTERVENTIONS:
Other: Dual Task Training — Exercise which combines cognitive task with motor task e.g Backward counting during sit ups.
  Calculation questions during stationary cycle for 10 mins. Sequentially perform movements on commands like normal standing (bipedal support with feet separated at shoulder width, Feet together (bipedal support with feet side by side), Semitandem stance, Tandem stance, one leg support on the dominant leg, one leg support on the nondominant leg by first laterally moving the trunk with shoulder abducted at least above 60 degree
  Other Names: Cognitive task + Motor Task
  Arms: Dual Task Training
Other: Task Specific Training — Wide based gait training.
  Auditory forward digit span:
  Remember as many as possible of the number/letter forward sequence, you were told
  Auditory backward digit span:
  Remember as many as possible of the number/letter back sequence, you were told
  Visual forward digit span:
  Remember as many as possible of the number forward sequence shown to you by means of cardboard
  Visual backward digit span:
  Remember as many as possible
  Other Names: cognitive task and motor task
  Arms: Task Specific Training

SUMMARY:
This study focuses on Dual Task Training as daily living involves many dual task conditions, in which a person requires to do two or more tasks at same time. without the ability to carry out these types of Dual movements. This study aims to improve the ability to do two tasks at same time, targeted to decrease the risk of fall in stroke patients. This study helps in understanding how multiple tasks simultaneously affects patients' abilities and creating effectiveness programs.

DETAILED DESCRIPTION:
The World Health Organization (WHO) defines the stroke as a brain injury that causes rapid and noticeable changes in cerebral function, lasting 24 hours or longer, or resulting in death. Strokes can be caused by vascular issues and include cerebral infarction, intracerebral hemorrhage, and subarachnoid hemorrhage. Stroke is a syndrome characterized by acute neurological deficits caused by vascular injury in the central nervous system. It's a major cause of disability and mortality globally, resulting from various risk factors, diseases, and mechanisms. Dual-task training refers to the ability to simultaneously perform multiple cognitive and motor activities while maintaining postural control. Divided attention is the capacity to do more than one thing at the same time. Dual-task training innovatively combines motor and cognitive rehabilitation in a comprehensive module. TST, or task-specific training, is a popular rehab approach that emphasizes function and is commonly used for stroke patients. It's all about targeting specific tasks to help with recovery.

RCT conducted on two groups, Dual Task Training and Task Specific training. interventions applied with a frequency of three times a week for eight weeks protocol. Participants will be divided into 2 groups. 1st group will receive Dual task training for motor and cognition simultaneously. 2nd group will receive task specific training for motor and cognition functioning.

ELIGIBILITY:
Inclusion Criteria:

* Patients with age ≥ 45 years' old both male and female.
* Patients with Mild cognitive impairment with MOCA score of 18-25.
* Patients with sub-acute or chronic stage of stroke and are able to sit
* independently for 30 secs.
* Patients with primary level education.

Exclusion Criteria:

* Patients with dementia that had been diagnosed by a neurologist.
* Patients with neurological, psychiatric, or medical disorders.
* Patients with auditory or visual impairments.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2024-05-30 (Actual); Primary Completion 2024-11-05 (Estimated); Study Completion 2024-12-05 (Estimated)

PRIMARY OUTCOMES:
Fugl Meyer Assessment Tool | 8th week
  The Fugyl-Meyer scale was developed as the first quantitative evaluative instrument for measuring sensorimotor stroke recovery.
Trail Making Test A and B | 8 weeks
  The Trail Making Test (TMT) is one of the most popular neuropsychological tests and is included in most test batteries.

SECONDARY OUTCOMES:
Digit Span Test | 8 weeks
  The Digit Sequencing or Digit Span test is one of the main tools developed to measure one's verbal working memory The Digit Sequence test is one of the main tools developed to measure one's verbal working memory, overall intelligence, attention, and cognitive functioning
stroop color and word test | 8 weeks
  The Stroop Color and Word Test (SCWT) is a neuropsychological test extensively used to assess the ability to inhibit cognitive interference that occurs when the processing of a specific stimulus feature impedes the simultaneous processing of a second stimulus attribute, well-known as the Stroop Effect
Modified Functional Reach Test | 8 weeks
  The Modified Functional Reach Test (MFRT) is a simple and adaptive clinical assessment instrument for determining sitting balance, an important part of functional ability.

CONTACTS AND LOCATIONS:
Overall Officials: Bushra Sultana, MSPT, Principal Investigator — Riphah International University
Locations (1):
- National Institute of Rehabilitation sciences, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Murphy SJ, Werring DJ. Stroke: causes and clinical features. Medicine (Abingdon). 2020 Sep;48(9):561-566. doi: 10.1016/j.mpmed.2020.06.002. Epub 2020 Aug 6. PMID 32837228
- [Background] Yeh TT, Chang KC, Wang JJ, Lin WC, Wu CY. Neuroplastic Changes Associated With Hybrid Exercise-Cognitive Training in Stroke Survivors With Mild Cognitive Decline: A Randomized Controlled Trial. Neurorehabil Neural Repair. 2023 Sep;37(9):662-673. doi: 10.1177/15459683231200220. PMID 37750660
- [Background] Feigin VL, Brainin M, Norrving B, Martins S, Sacco RL, Hacke W, Fisher M, Pandian J, Lindsay P. World Stroke Organization (WSO): Global Stroke Fact Sheet 2022. Int J Stroke. 2022 Jan;17(1):18-29. doi: 10.1177/17474930211065917. PMID 34986727
- [Background] Wolfe CD. The impact of stroke. Br Med Bull. 2000;56(2):275-86. doi: 10.1258/0007142001903120. PMID 11092079
- [Background] Langhorne P, Bernhardt J, Kwakkel G. Stroke rehabilitation. Lancet. 2011 May 14;377(9778):1693-702. doi: 10.1016/S0140-6736(11)60325-5. PMID 21571152
- [Background] Rost NS, Brodtmann A, Pase MP, van Veluw SJ, Biffi A, Duering M, Hinman JD, Dichgans M. Post-Stroke Cognitive Impairment and Dementia. Circ Res. 2022 Apr 15;130(8):1252-1271. doi: 10.1161/CIRCRESAHA.122.319951. Epub 2022 Apr 14. PMID 35420911
- [Background] Traxler K, Schinabeck F, Baum E, Klotz E, Seebacher B. Feasibility of a specific task-oriented training versus its combination with manual therapy on balance and mobility in people post stroke at the chronic stage: study protocol for a pilot randomised controlled trial. Pilot Feasibility Stud. 2021 Jul 27;7(1):146. doi: 10.1186/s40814-021-00886-0. PMID 34311772
- [Background] V.Rajalaxmi JA. Effects of Dual Task Training Versus PNF Pattern on Balance and Cognition in geriatrics population. International Journal of Life science and Pharma Research. 2022 July; 12(4).
- [Background] Xiao Y, Yang T, Shang H. The Impact of Motor-Cognitive Dual-Task Training on Physical and Cognitive Functions in Parkinson's Disease. Brain Sci. 2023 Mar 3;13(3):437. doi: 10.3390/brainsci13030437. PMID 36979247
- [Background] Kim KH, Jang SH. Effects of Task-Specific Training after Cognitive Sensorimotor Exercise on Proprioception, Spasticity, and Gait Speed in Stroke Patients: A Randomized Controlled Study. Medicina (Kaunas). 2021 Oct 13;57(10):1098. doi: 10.3390/medicina57101098. PMID 34684135
- [Background] Iqbal M, Arsh A, Hammad SM, Haq IU, Darain H. Comparison of dual task specific training and conventional physical therapy in ambulation of hemiplegic stroke patients: A randomized controlled trial. J Pak Med Assoc. 2020 Jan;70(1):7-10. doi: 10.47391/JPMA.10443. PMID 31954014
- [Background] Kim H Yeh. Reliability, concurrent validity, and responsiveness of the FuglMeyer Assessment (FMA) for hemiplegic patients. Journal Of Physical Therapy Science. 2012; 24(9): 893.
- [Background] Marchesi G, Ballardini G, Barone L, Giannoni P, Lentino C, De Luca A, Casadio M. Modified Functional Reach Test: Upper-Body Kinematics and Muscular Activity in Chronic Stroke Survivors. Sensors (Basel). 2021 Dec 29;22(1):230. doi: 10.3390/s22010230. PMID 35009772
- [Background] Katz-Leurer M, Fisher I, Neeb M, Schwartz I, Carmeli E. Reliability and validity of the modified functional reach test at the sub-acute stage post-stroke. Disabil Rehabil. 2009;31(3):243-8. doi: 10.1080/09638280801927830. PMID 18608433
- [Background] Lam B, Middleton LE, Masellis M, Stuss DT, Harry RD, Kiss A, Black SE. Criterion and convergent validity of the Montreal cognitive assessment with screening and standardized neuropsychological testing. J Am Geriatr Soc. 2013 Dec;61(12):2181-2185. doi: 10.1111/jgs.12541. Epub 2013 Dec 9. PMID 24320735
- [Background] Tombaugh TN. Trail Making Test A and B: normative data stratified by age and education. Arch Clin Neuropsychol. 2004 Mar;19(2):203-14. doi: 10.1016/S0887-6177(03)00039-8. PMID 15010086
- [Background] Muangpaisan W, Intalapaporn S, Assantachai P. Digit span and verbal fluency tests in patients with mild cognitive impairment and normal subjects in Thai-community. J Med Assoc Thai. 2010 Feb;93(2):224-30. PMID 20302005
- [Background] Scarpina F, Tagini S. The Stroop Color and Word Test. Front Psychol. 2017 Apr 12;8:557. doi: 10.3389/fpsyg.2017.00557. eCollection 2017. PMID 28446889